CLINICAL TRIAL: NCT02557269
Title: Real Life Proof-of-Concept Study to Assess the Effect of Methylcellulose as add-on "Seal" to the In-season Pharmacologic Rescue Treatment in Subjects With Allergic Rhinitis
Brief Title: 4"S" - Seasonal Symptoms Suppression Study
Acronym: 4"S"
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association Asthma, Bulgaria (Other)
Collaborators: Nasaleze (Industry)
Responsible Party: Principal Investigator, Prof. Todor Popov, Professor, Association Asthma, Bulgaria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSSS2015
Record Dates: First submitted 2015-07-17; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Pollenosis; Congestion; Mucoadhesive Treatment; Nasal Decongestant; Nasal Antihistamine; Nasal Corticosteroid
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Mometasone Furoate; bilastine; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group HPMC (Active Comparator): Hydroxyl-propyl-methyl-cellulose (HPMC) powder added immediately after other intranasal treatment options
  Interventions: Drug: Xylometazoline - intranasal application; Drug: Azelastine - intranasal application; Drug: Mometasone furoate - intranasal application; Drug: Hydroxyl-propyl-methyl cellulose powder - intranasal application; Drug: Bilastine 20 mg; Drug: Prednisolone 5 mg
- Group Placebo (Placebo Comparator): Lactose powder (placebo) added immediately after other intranasal treatment options
  Interventions: Drug: Xylometazoline - intranasal application; Drug: Azelastine - intranasal application; Drug: Mometasone furoate - intranasal application; Other: Placebo - Lactose powder; Drug: Bilastine 20 mg; Drug: Prednisolone 5 mg
- Group Immunotherapy (Other): Immunotherapy group with grass allergens sublingually (Staloral #688) and rescue medication
  Interventions: Drug: Xylometazoline - intranasal application; Drug: Azelastine - intranasal application; Drug: Mometasone furoate - intranasal application; Drug: Bilastine 20 mg; Drug: Prednisolone 5 mg

INTERVENTIONS:
Drug: Xylometazoline - intranasal application — Applied as needed up to 5 consecutive days when prominent congestion
Drug: Azelastine - intranasal application — Applied as needed when prominent symptom is rhinorrhea
  Other Names: Allergodil
Drug: Mometasone furoate - intranasal application — Applied once daily (2 puffs) when no satisfactory therapeutic control from other intranasal treatment
  Other Names: Nasonex
Drug: Hydroxyl-propyl-methyl cellulose powder - intranasal application — Applied intranasally immediately after every application other intranasal formulation
  Other Names: Nasaleze
  Arms: Group HPMC
Other: Placebo - Lactose powder — Applied intranasally immediately after every application other intranasal formulation
  Arms: Group Placebo
Drug: Bilastine 20 mg — 1 tablet per os - as needed
  Other Names: Fortecal
Drug: Prednisolone 5 mg — Per os - if needed (only in case of broncial obstruction)

SUMMARY:
ASIT naïve patients sensitized to grass pollens will be recruited for the study. All of them will be instructed to treat bothersome in-season symptoms when they appear (on as needed, pro re nata basis) with rescue medication. They will be given 5 different options and will be informed about the effects of each of them in order to make their optimal choice for different symptoms and their combination: local decongestant (xylomethazoline, when congestion is leading), local antihistamine (azelastine, when itching, sneezing and rhinorhea a predominant), nasal corticosteroid (momethasone, when all nasal symptoms are pressing and no adequate relief is obtained form the other 2 local treatments), oral antihistamine (bilastine, when itching and sneezing persist despite the local treatments) and oral corticosteroid (prednisolone, when any or all symptoms become unbearable despite the other suggested treatments). Patients who are reluctant to use immunotherapy or who are too late to initiate it will be randomized to be treated with the listed medications on as needed basis, the nasally applied formulations will be followed by either HPMC to prolong and enhance their effect (Group HPMC) or placebo (lactose powder) (Group Placebo) to serve as control. Patients indicated and willing to carry out ASIT will be treated according to the standard protocol with grass allergens sublingually (Staloral #688) and will receive rescue medication (Group Immunotherapy).

DETAILED DESCRIPTION:
Rationale. Assessment and follow up of specifically sensitized subjects with allergic rhinitis during the pollen season is traditionally based on symptom scores. Accounting for the use of rescue medication on top of symptom scores provides another dimension to the overall clinical characterization of the patients. Thus, using "combined symptom and medication scores" (CSMS) allows thorough characterization of the disease course. Guidelines recommend that CSMS are used for assessment of the effect of allergen specific immunotherapy in subjects with allergic rhinitis. Different allergic rhinitis management strategies can be evaluated and compared by means of CSMS. In the update of the ARIA guidelines of 2010, 24 recommendations have been made in relation to pharmacologic treatment. Special position paper has been devoted to severe chronic upper airway disease (SCUAD), the treatment for which has been earmarked as unmet need.

Consequently, a standardized and universally recognized rescue treatment strategy does not exist. The most common approach for handling nasal complaints in real life consists in using rescue medication for symptoms whenever they appear. This is certainly the case when symptoms appear for the first time ever, or when patients do not want to resort to allergen specific immunotherapy (ASIT) and / or regular oral antihistamine treatment for financial reasons or personal beliefs. Under these circumstances, a long list of pharmacological choices for local or systemic application is possible including antihistamines, corticosteroids, leukotriene antagonists, cromones and antimuscarinic drugs.

Formulations for local application in the nose appeal to patients with their ease of use and immediate relief. They comprise a variety of generic drugs: decongestants, antihistamines, corticosteroids and antimuscarinics. The fact that they are not ingested makes them first choice for people reluctant to take oral medications. In many cases it is possible to control the symptoms of allergic rhinitis with these formulations used per se or as adjunct rescue medication in the course of ASIT.

The question stays whether the effectiveness of nasally applied drugs can further be improved. Despite the good rationale for their mechanism of action, their efficacy is diminished by the cleaning mechanisms of the nose, rhinorrhea in particular. Slowing down of the clearance of the nasal mucosa and prolonging the contact time with the nasal mucosa would enhance their pharmaceutical effects. The investigators have demonstrated by objectively measuring nasal flow rates that "sealing" in place locally applied oxymetazoline in subjects with persistent allergic rhinitis by means of commercially available hydroxyl-propyl-methyl-cellulose (HPMC) significantly enhances the resulting decongestion and that this effect is augmented over a time span of 2 weeks without noticeable tachyphylaxis or adverse events.

The investigators set the aim to investigate whether this beneficial effect of HPMC translates into clinical benefits in a real life clinical trial for other available drug preparations for nasal delivery.

Study design. ASIT naïve patients sensitized to grass pollens will be recruited for the study. All of the patients will be instructed to treat bothersome in-season symptoms when they appear (on as needed, pro re nata basis) with rescue medication. The patients will be given 5 different options and will be informed about the effects of each of them in order to make their optimal choice for different symptoms and their combination: local decongestant (xylomethazoline, when congestion is leading), local antihistamine (azelastine, when itching, sneezing and rhinorhea a predominant), nasal corticosteroid (momethasone, when all nasal symptoms are pressing and no adequate relief is obtained form the other 2 local treatments), oral antihistamine (bilastine, when itching and sneezing persist despite the local treatments) and oral corticosteroid (prednisolone, when any or all symptoms become unbearable despite the other suggested treatments). Patients who are reluctant to use immunotherapy or who are too late to initiate it will be randomized to be treated with the listed medications on as needed basis, the nasally applied formulations will be followed by either HPMC to prolong and enhance their effect (Group HPMC) or placebo (lactose powder) (Group Placebo) to serve as control. Patients indicated and willing to carry out ASIT will be treated according to the standard protocol with grass allergens sublingually (Staloral #688) and will receive rescue medication (Group Immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Age ≥ 18 and ≤ 55 years
* Personal history of rhinitis during the pollen season
* Moderately severe / severe seasonal allergic rhinitis (grass)
* Positive skin prick test for grass/cereals

Exclusion Criteria:

* Subjects with arterial hypertension, arrhythmia or evidence of heart ischemia
* Subjects with other serious chronic comorbidities and bad therapeutic control
* Subjects with nasal polyposis
* Any contraindications for xylometazoline
* Any contraindications for HPMC
* Any contraindications for azelastine
* Any contraindications for bilastine
* Any contraindications for mometasone
* Any contraindications for prednisolone
* Subjects unable to give informed consent
* Pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Combined Sypmtom and Medication Score | Up to 6 months
  The primary outcome will be comparison of total combined symptoms and medication scores (TCSMS) collected from patients' diaries for a fixed period during the pollen season

SECONDARY OUTCOMES:
Drug Specific Combined Sypmtom and Medication Score | Up to 6 months
  Drug specific combined symptoms and medication scores (DsCSMS) will be calculated for each rescue medication and compared between the 3 arms of the trial.
Visual Analogue Scale | Up to 6 months
  Visual analogue scale (VAS) scores (Scores range from 0 [no symptoms] to 10 [worst possible symptoms]) at each visit and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Todor A Popov, MD, PhD, Principal Investigator — Medical University of Sofia
Locations (1):
- Medical University Sofia, University Hospital "Alexandrovska", Clinic of Allergy and Asthma, Sofia, Bulgaria

REFERENCES:
- [Background] Pfaar O, Demoly P, Gerth van Wijk R, Bonini S, Bousquet J, Canonica GW, Durham SR, Jacobsen L, Malling HJ, Mosges R, Papadopoulos NG, Rak S, Rodriguez del Rio P, Valovirta E, Wahn U, Calderon MA; European Academy of Allergy and Clinical Immunology. Recommendations for the standardization of clinical outcomes used in allergen immunotherapy trials for allergic rhinoconjunctivitis: an EAACI Position Paper. Allergy. 2014 Jul;69(7):854-67. doi: 10.1111/all.12383. Epub 2014 Apr 25. PMID 24761804
- [Background] Calderon MA, Bernstein DI, Blaiss M, Andersen JS, Nolte H. A comparative analysis of symptom and medication scoring methods used in clinical trials of sublingual immunotherapy for seasonal allergic rhinitis. Clin Exp Allergy. 2014 Oct;44(10):1228-39. doi: 10.1111/cea.12331. PMID 24773171
- [Background] Brozek JL, Bousquet J, Baena-Cagnani CE, Bonini S, Canonica GW, Casale TB, van Wijk RG, Ohta K, Zuberbier T, Schunemann HJ; Global Allergy and Asthma European Network; Grading of Recommendations Assessment, Development and Evaluation Working Group. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines: 2010 revision. J Allergy Clin Immunol. 2010 Sep;126(3):466-76. doi: 10.1016/j.jaci.2010.06.047. PMID 20816182
- [Background] Bousquet J, Bachert C, Canonica GW, Casale TB, Cruz AA, Lockey RJ, Zuberbier T; Extended Global Allergy and Asthma European Network, World Allergy Organization and Allergic Rhinitis and its Impact on Asthma Study Group. Unmet needs in severe chronic upper airway disease (SCUAD). J Allergy Clin Immunol. 2009 Sep;124(3):428-33. doi: 10.1016/j.jaci.2009.06.027. Epub 2009 Aug 5. PMID 19660803
- [Background] Valerieva A, Popov TA, Staevska M, Kralimarkova T, Petkova E, Valerieva E, Mustakov T, Lazarova T, Dimitrov V, Church MK. Effect of micronized cellulose powder on the efficacy of topical oxymetazoline in allergic rhinitis. Allergy Asthma Proc. 2015 Nov-Dec;36(6):e134-9. doi: 10.2500/aap.2015.36.3879. Epub 2015 Jun 29. PMID 26133030